CLINICAL TRIAL: NCT00598494
Title: Effect of Bedrest With and Without Exercise on Cardiac Atrophy: Synergistic Supplemental Testing With the Cleveland Clinic Bedrest Study
Brief Title: Effect of Bedrest With and Without Exercise on the Heart
Status: Terminated | Type: Observational
Why Stopped: Main bedrest study moved to Texas. No enrollment at Cleveland Clinic.
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Space Biomedical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 07-007; SMS00404 (Other Grant/Funding Number: NSBRI)
Record Dates: First submitted 2007-12-26; First posted 2008-01-22 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Bedrest
Keywords: effect of bedrest; cardiac atrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research sub-study is to determine the changes in heart function during the bedrest period using ultrasound and MRI. This topic is important for medical care of astronauts in space. It can enable physicians on the ground to monitor exercise protocols that are used to prevent deconditioning-loss of strength during long space flights.

Your participation in this study would include ultrasound examinations with bicycle exercise before, during, and after the 12-week bedrest period. MRI exams would be performed before and after the bedrest period.

Each echo exam may last up to 1 hour. This time will be required to perform an ultrasound examination before and during supine (lying down) bicycle exercise. The exercise period will be approximately 10-15 minutes. The bicycle exercise will be a symptom-limited test. This means that the test will be stopped if you experience any discomfort. An ultrasound examination of your heart will be done to assess heart function. You will be asked to lie on your left side on an examination table while a technician takes pictures of your heart with a small probe that is gently pressed against your chest after applying a gel. The ultrasound data will be processed to evaluate myocardial strain, a value that may be useful in describing heart function.

Each MRI may last up to 1 hour. An MRI obtains body pictures created by using magnetic energy rather than x-ray energy. To have the scan, you will lie on a table that slides into the scanner, which is like a large tube. An MRI examination of your heart will be done to assess heart function. You will be asked to lie still and follow simple breathing instructions during the procedure. The MRI data will be processed to evaluate the volume of blood being pumped by your heart, a value that may be useful in describing heart function.

DETAILED DESCRIPTION:
NASA and NSBRI are making considerable investment in a bedrest study being conducted at the Cleveland Clinic Foundation under the directorship of Peter Cavanaugh, primarily to assess the impact of exercise on prevention of osteoporosis in a twelve-week bedrest study to simulate microgravity. This provides an outstanding opportunity for synergistic add-on studies to combine the resources of the bone team of NSBRI with those of the Cardiovascular Alterations and Smart Medicine by conducting a series of detailed echocardiographic and computed tomographic examinations of the heart in these patients. These studies will serve to advance a number of the specific aims of a grant currently held by James D. Thomas from NSBRI concerning both the primary effects of microgravity on the heart and its reversal with exercise as well as the ability to prove out new echocardiographic methods for measuring the cardiac response to exercise. Finally, they will provide an excellent opportunity to prove out methodologies being developed for remote delivery of healthcare by image fusion from free-flight studies to in-flight echoes.

We will to pursue the following specific aims with this synergistic study:

Specific Aim 1: To assess the impact of bedrest on cardiac atrophy, stiffening of the left ventricular diastolic pressure volume curve, and exercise tolerance and ventricular mechanics and demonstrate at least partial prevention of these changes with the proposed exercise prescription.

Specific Aim 2: To demonstrate the ability of novel echocardiographic indices of ventricular function (strain, torsion, IVPG) to predict functional capacity and response to exercise.

Specific Aim 3: To test whether pre-bedrest MRI examinations could be co-registered with bedrest 3D echocardiographic exams to track atrophy and altered cardiac anatomy. The ability of detailed 3D ground examinations to be compared precisely with in-flight 3D echos is a key goal of autonomous medical care system for expedition class missions.

Proposed Protocol (summary):

Pre-bedrest (within 1-3 weeks prior):

1. Resting two and three-dimensional echocardiogram.
2. Maximal supine bicycle test with echocardiographic assessment of wall motion, tissue strain, tissue torsion, and intraventricular pressure gradients (IVPG) by color M-mode flow propagation. In addition to the peak exercise assessment, we will also focus on the submaximal level (heart rate ~100).
3. MRI examination of the heart for LV volume and mass and subsequent cross registration with echocardiogram.

Six weeks of bedrest:

1. Resting two and three-dimensional echo exam.
2. Low-level supine bicycle exercise echo (HR no greater than 100) with torsion, strain, and IVPG assessment.

Twelve weeks of bedrest:

1. Resting two and three-dimensional echo.
2. Maximal supine bicycle test with echocardiographic assessment of wall motion, tissue strain, tissue torsion, and IVPG.
3. MRI examination of the heart.

As part of the overall bedrest protocol (IRB 6504), patients will be randomized either to complete bedrest with negative tilt vs. those who will undergo daily horizontal treadmill exercise to replace the calcaneus impact measured pre-bedrest in the same subjects. This provides an excellent opportunity for assessing the impact of this degree in type of exercise on the cardiovascular system.

The specific aims of this synergistic study will be answered as follows:

Specific Aim 1: To assess the impact of bedrest on cardiac atrophy, stiffening of the left ventricular diastolic pressure volume curve, and exercise tolerance and ventricular mechanics and demonstrate at least partial prevention of these changes with the proposed exercise prescription.

LV mass will be measured by MRI pre- and post-bedrest and by 3D echo at bedrest stages. Two-way linear regression will be used to determine change over time in LV mass and to compare the response to exercise. Similarly, exercise capacity will be analyzed. Among the LV mechanics parameters that will be available for analysis at all 3 data acquisition points are: (resting) LV end-diastolic and end-systolic volume, left atrial volume, transmitral E and A waves and E-wave deceleration time, Doppler tissue annular E, A, and S waves, radial, circumferential, and longitudinal strain at the midventricular level, LV torsion and peak untwisting rate, and color M-mode IVPG. These same parameters will also be available for analysis during low-level (HR 100) bicycle exercise.

Specific Aim 2: To demonstrate the ability of novel echocardiographic indices of ventricular function at rest (strain, torsion, IVPG) to predict functional capacity and response to exercise.

Strain, torsion, and IVPG will be assessed at all stages and correlated with changes in cardiac atrophy parameters (LV mass and volumes).

Specific Aim 3: To test whether pre/post bedrest MRI examinations can be co-registered with bedrest 3D echocardiographic exams to track atrophy and altered cardiac anatomy. The ability of detailed 3D ground examinations to be compared precisely with in-flight 3D echos is a key goal of autonomous medical care system for expedition class missions.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* Currently participating in bed rest study

Exclusion Criteria

-unable to maintain bedrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal volunteers
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2007-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
2D and 3D echocardiography | 12 weeks

SECONDARY OUTCOMES:
MRI | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jim Thomas, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No